CLINICAL TRIAL: NCT01977963
Title: Genetic Study of Antithyroid Drugs Associated Agranulocytosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201112083RID
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-10

CONDITIONS: Agranulocytosis
MeSH Terms: conditions — Agranulocytosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Agranulocytosis

SUMMARY:
Thionamides, the antithyroid drugs, have been widely used to treat hyperthyroidism1. Side effects are found in 1% - 5% of the patients1. One of the most serious side effect is agranulocytosis, which occurs in 0.1% - 0.3 % of the patients1. This might lead to severe infection and sometimes mortality. The underlying mechanism is unclear. An immune phenomenon may be involved because the antigranulocyte antibodies or lymphocyte sensitized to antithyroid drugs are found in these patients6,7. The recognition of major histocompatibility complex class II peptide complexes by T lymphocytes is central to the development of immune response. According to a report in 1996, the HLA DRB1*08032 allele is strongly associated with susceptibility to methimazole-induced agranulocytosis20.

Recently, there are new techniques for genetics study. We aimed to identify the associated genetic change of the agranulocytosis side effect of antithyroid drugs. First, we will look at the classical human Leukocyte Antigen (HLA) loci, such as HLA-A, -B, -C, -DR, -DQ and -DP. If no significant change is found in the above genes, we will consider whole exon sequencing with next-generation sequencing, Statistic analysis will include appropriate linkage analysis, association study, variation data analysis, pathway analysis. If we can identify the genetic change and perform genetic examinations before prescription, we can avoid the happening of severe side effects.

ELIGIBILITY:
Inclusion Criteria:

* patients with absolute neutrophil count lower than 500/mm3 caused by anti-thyroid drugs

Exclusion Criteria:

* Patients who is younger than 20 years old or older than 85 years old

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Agranulocytosis caused by anti-thyroid drugs
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-04; Primary Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with anti-thyroid drug related agranulocytosis | within 2 month after taking the drug
  The investigators review the chart to see if the patients had anti-thyroid drug related agranulocytosis

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan